CLINICAL TRIAL: NCT05831800
Title: Assessing Hydration Status With a Wearable Bioimpedance Sensor in Elderly Individuals - A Prospective Feasibility Study
Brief Title: Assessing Hydration Status With a Wearable Bioimpedance Sensor in Elderly Individuals
Acronym: HELD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mode Sensors AS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CTR0061A HELD
Record Dates: First submitted 2023-03-27; First posted 2023-04-26 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Dehydration
MeSH Terms: conditions — Dehydration

STUDY DESIGN:
Intervention Model Description: Single-arm prospective feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Wearable bioimpedance sensor (Other)
  Interventions: Device: Wearable bioimpedance sensor

INTERVENTIONS:
Device: Wearable bioimpedance sensor — The investigational device is an electronic bioimpedance-based, body-worn, battery-powered sensor intended to monitor changes in fluid balance. It is designed as an adhesive patch with four integrated electrodes. The outer electrodes are used to supply a low current, while the inner electrodes are used for voltage measurements.

SUMMARY:
This is a single-arm prospective study, investigating the feasibility, usability, and safety of a wearable bioimpedance sensor in elderly individuals. The sensor is applied on the upper back of the subject, and will be replaced once weekly. The study will include four phases, each interspersed by an interim analysis. Each phase will have a duration of four weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years

Exclusion Criteria:

* Known allergies or skin sensitivities to electrode hydrogel and/or acrylic-based adhesives
* Non-intact skin such as skin breakdown where the device is to be placed (upper back)
* Implantable pulse generators such as pacemakers and defibrillators
* Any medical or psychiatric condition, which in the opinion of the investigator precludes participation

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-06-14 (Actual); Primary Completion 2024-12-20 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Mean use time of the wearable sensor | Up to 7 days

SECONDARY OUTCOMES:
The mean number of days the sensor provides valid measurements | Up to 7 days
Mean and standard deviation of the device output variables | Up to 7 days
Stability of device measurements following weekly patch replacement | Day 8, 15, 22, 29
  Test-retest reliability of the investigational device will be investigated by assessing the correlation between impedance measurements (in Ohm) before and after device replacement.
Clinical assessment of hydration status | Day 1, 8, 15, 22, 29
User satisfaction | Day 8, 15, 22, 29
  Will be assessed using a likert scale from 1-5, where 1 represents "strongly disagree" and 5 represents "strongly agree".
Frequency and severity of adverse device effects | Day 1-30

CONTACTS AND LOCATIONS:
Overall Officials: Sigve N Aas, PhD, Study Director — Mode Sensors AS
Locations (1):
- Tempe Helse- og velferdssenter, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No